CLINICAL TRIAL: NCT01346384
Title: Time - Related Cuff Pressure and Volume of the Laryngeal Tube With the Use of Nitrous Oxide
Status: Completed | Type: Observational
Sponsor: Prince of Songkla University (Other)
Responsible Party: Assistant Professor Nalinee Kovitwanawong, Department of Anesthesiology Faculty of Medicine Prince of Songkla University Thailand
Other Study IDs: LT-N2O
Record Dates: First submitted 2011-04-25; First posted 2011-05-03 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-04

CONDITIONS: Adult Disease
Keywords: intracuff pressure; laryngeal tube; nitrous oxide
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- intracuff pressure N2O: measured intracuff pressure of LT with N2o during operative period
  Interventions: Device: laryngeal tube (VBM Medizintechnik)

INTERVENTIONS:
Device: laryngeal tube (VBM Medizintechnik) — laryngeal tube number 4
  Other Names: The laryngeal tube (VBM Medizintechnik, Sulz, Germany)

SUMMARY:
The purpose of this study is to investigate the time-related intracuff pressure and volume change (which reflects the pharyngeal pressure) of the LT during anesthesia with N2O.

DETAILED DESCRIPTION:
Background : The laryngeal tube airway (LT) is an extraglottic airway device with a proximal and distal conical cuff designed to secure a patient's airway during either spontaneous breathing or controlled ventilation. Application of this device with the use of N2O may be related to the ischemic change of the oropharyngeal mucosa. The objective of this study was to investigate the time-related intracuff pressure and volume change (which reflects the pharyngeal pressure) of the LT during anesthesia with N2O.

Methods : Seventy-five patients were studied with the use of LT size 4. N2O (66%) and isoflurane were used to maintain anesthesia. Initial intracuff pressure and volume were recorded for airway sealing during ventilation. Time-course changes of the intracuff pressure followed by recording every 10 min. If the intracuff pressure reached 100 cmH2O, the cuff was deflated to the initial intracuff pressure and the volume of deflated air and postoperative airway complications were recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist physical status I or II
* Undergoing elective orthopedic surgery and surgery of breast under general anesthesia with an expected duration of 60 min or more

Exclusion Criteria:

* Height was < 155 or >180 cm (for the use of laryngeal tube size 4)
* Body mass index ≥35 kg/m2
* Preexisting laryngotracheal disease
* Risk of pulmonary aspiration of gastric contents.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
intracuff pressure | 1-4 hours
  measured intracuff pressure of LT with N2O during intraoperative period

CONTACTS AND LOCATIONS:
Locations (1):
- Songklanagarind Hospital, Hat Yai, Changwat Songkhla, Thailand